CLINICAL TRIAL: NCT04928586
Title: Efficacy, Safety and Predictive Indicators of Immunosuppressant Combined With Pirfenidone in the Treatment of Connective Tissue Disease-related Interstitial Lung Disease (CTD-ILD)
Brief Title: Immunosuppressant Combined With Pirfenidone in CTD-ILD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTD-ILD QiluH
Record Dates: First submitted 2021-05-27; First posted 2021-06-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pirfenidone; Connective Tissue Diseases; Interstitial Lung Disease
Keywords: pirfenidone; interstitial lung disease; connective tissue disease; rheumatoid arthritis; systemic sclerosis; inflammatory myopathy
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Arthritis, Rheumatoid; Scleroderma, Systemic; Myositis | interventions — pirfenidone; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pirfenidone group (Experimental): CTD-ILD patients treated with DMARDs and pirfenidone
  Interventions: Drug: Pirfenidone; Drug: DMARDs
- No-Pirfenidone group (Active Comparator): CTD-ILD patients treated with DMARDs, without pirfenidone
  Interventions: Drug: DMARDs

INTERVENTIONS:
Drug: Pirfenidone — CTD-ILD patients treated with pirfenidone up to the maximum tolerable dose
  Arms: Pirfenidone group
Drug: DMARDs — CTD-ILD patients treated with DMARDs according to the condition of the disease

SUMMARY:
A prospective cohort study was used to observe the efficacy and safety of different immunosuppressive agents with/wo pirfenidone on CTD-ILD patients in Qilu Hospital of Shandong University for 36 months.The main research endpoints are lung function, patient dyspnea score, 6-minute walking distance, imaging indicators, primary disease activity, adverse reactions, etc.

DETAILED DESCRIPTION:
This study will enroll 200 cases of connective tissue disease-related interstitial lung disease (CTD-ILD) patients in China, including inflammatory myopathy (IIM) patients, rheumatoid arthritis (RA) patients, systemic sclerosis (SSc) patients, Sjogren's syndrome (SS) patients and other connective tissue disease patients.According to the patient's condition,the participants plan to be treated with different immunosuppressive agents with/wo pirfenidone .Participants can choose to continue the study up to 36 months.The efficacy and safety of the treatment in CTD-ILD patients will be evaluated with lung function, quality of life / cardiopulmonary function assessment and other disease activity indices.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the following inclusion criteria will be eligible to participate in the study:

  1. Aged 18-80 years;
  2. In accordance with the diagnostic criteria of connective tissue disease-related pulmonary interstitial disease (CTD-ILD);The diagnosis of CTD is in line with the international classification standard of rheumatism (including inflammatory myopathy, systemic sclerosis, rheumatoid arthritis, sjogren's syndrome, systemic lupus erythematosus, mixed connective tissue disease, undifferentiated connective tissue disease);
  3. Subjects are willing to participate and use medication and follow-up time according to the treatment plan, and sign the informed consent;

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study:

  1. Subjects have non-diffuse connective tissue disease or other arthritis other than RA, such as ANCA-relateed vasculitis, psoriatic arthritis, etc;
  2. Patients who have ILD with clear etiology, such as HIV, GVHD ；
  3. Combined viscera function significantly abnormal patient:

     1. Liver: AST, ALT >1.3ULN; Bilirubin >1.5 ULN; or previous diagnosis of viral hepatitis;
     2. Kidney: Creatinine clearance <30 mL/min;
     3. Lung: Airway obstruction (pre-bronchodilator FEV1/FVC <0.7); pleural effusion accounts for more than 20% of pleural effusion ;severe pulmonary infection or other clinically significant pulmonary abnormalities;
     4. Cardiovascular: Myocardial infarction or unstable angina within six months;
     5. Gastrointestinal tract: With active peptic ulcer or bleeding;
     6. Blood system: Severe anemia, decreased white blood cells and platelets
     7. Nervous system: Patients with mental disorders; cerebral thrombosis events within the past 1 year;
  4. Combined with poor prognosis of diseases, such as cancer, genetic diseases and so on;
  5. Women during pregnancy or lactation or childbearing age cannot ensure effective contraception;
  6. According to the researchers, exhibited evidence of alcohol or drug abuse;
  7. Any other major medical events beyond control;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in FVC | 12 months
  Change in forced vital capacity(FVC) from 12 months to baseline
Change in DLCo | 12 months
  Change in carbon monoxide diffusing capacity (DLCo) from 12 months to baseline

SECONDARY OUTCOMES:
Changes in FVC | 6 months，24 months，36 months
  Changes from baseline in forced vital capacity(FVC)
Changes in DLCo | 6 months，24 months，36 months
  Changes from baseline in carbon monoxide diffusing capacity (DLCo)
Changes from baseline in Dyspnea score | 6 months，12 months, 24 months，36 months
  Changes from baseline in Dyspnea score. Dyspnea score:activity tolerance of patients with dyspnea in daily life: 0: normal, 1: dyspnea when climbing the fifth floor, 2: dyspnea when climbing the third floor, 3: dyspnea when climbing the second floor, 4: Difficulty in breathing when walking on the flat ground 100-500m, 5: Difficulty in breathing when walking on flat ground for 50-100m, 6: Difficulty in breathing when walking on flat ground for 15-50m, 7: Difficulty in breathing when walking on flat ground 5-15m, 8: Difficulty in breathing during daily dressing, 9: Difficulty in breathing when eating, 10: Difficulty in breathing when resting.The higher the score, the more severe the disease.
Imaging changes | 6 months，12 months, 24 months，36 months
  Changes from baseline in high-resolution computed tomography (HRCT)
Changes from baseline in 6 minutes walking distance | 6 months，12 months, 24 months，36 months
  Changes from baseline in 6 minutes walking distance
Changes from baseline in C-reactive protein(CRP) | 6 months，12 months, 24 months，36 months
  Changes from baseline in C-reactive protein(CRP)
Changes from baseline in Erythrocyte Sedimentation Rate(ESR) | 6 months，12 months, 24 months，36 months
  Changes from baseline in Erythrocyte Sedimentation Rate(ESR)
Changes from baseline in VAS score | 6 months，12 months, 24 months，36 months
  The visual analogue scale (VAS) is used for pain assessment. The basic method is to use a moving ruler with a length of about 10cm. One side is marked with 10 scales. The two ends are respectively "0" and "10" points. A point of 0 means no pain, and a point of 10 means the most unbearable. Severe pain. It can reflect the degree of activity of the primary disease.
Number of participants with "adverse events (AEs)" | Up to month 36
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiaoyun, Dr., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China